CLINICAL TRIAL: NCT00798993
Title: The Effect of 25-hydroxyvitamin D Supplementation and a Structured Exercise Program on Exercise Capacity and Quality of Life in Dialysis Patients
Brief Title: Effect of 25-hydroxyvitamin D and a Structured Exercise Program on Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Charles Gairdner Hospital (Other)
Responsible Party: Principal Investigator, Neil Boudville, Associate Professor, Sir Charles Gairdner Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCGH25OHD2008
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: End Stage Kidney Disease
Keywords: Chronic kidney failure; 25 hydroxyvitamin D; falls; exercise; quadriceps strength
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Cholecalciferol; 25-hydroxyvitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Structured exercise program (Active Comparator): Participants will be randomised at 3 months into either this group or the comparator of usual exercise.
  Interventions: Other: Structured Exercise program
- Vitamin D (Experimental): Cholecalciferol 2000U per day will be given to all participants for the duration of the study
  Interventions: Drug: Cholecalciferol (25-Hydroxyvitamin D)
- Usual exercise (Placebo Comparator): Participants randomised to this arm, at 3 months, will continue on their usual exercise routine
  Interventions: Other: Usual exercise

INTERVENTIONS:
Other: Structured Exercise program — 30 minutes on an exercise bicycle during every dialysis
  Arms: Structured exercise program
Drug: Cholecalciferol (25-Hydroxyvitamin D) — Cholecalciferol 2000U per day will be given for duration of study to all participants
  Arms: Vitamin D
Other: Usual exercise — Participants randomised to this arm at 3 months will continue on their usual exercise routine for the remaining 3 months
  Arms: Usual exercise

SUMMARY:
This study aims to examine the effect of 25 hydroxyvitamin D supplementation and a structured exercise program on the exercise capacity and quality of life of haemodialysis patients with 25 hydroxyvitamin D insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Stable on dialysis for at least 3 months
2. Able to obtain informed consent
3. Medically stable
4. Dialysis adequacy at target for small solute clearance (ie Kt/V>1.2 or Urea reduction ratio>65%)
5. Serum 25-hydroxyvitamin D levels less than 75nmol/L at baseline

Exclusion Criteria:

1. Limb Amputation
2. Impaired cognition
3. Impaired vision
4. Haemoglobin concentration < 110g/L
5. Change in Erythropoiesis stimulating agent dose over the last 2 months
6. Unable or unwilling to comply with exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Exercise capacity - modified shuttle walk test | Basesline, 3 & 6 months

SECONDARY OUTCOMES:
Quality of life with KDQOL | Baseline, 3 & 6 months
Quadriceps Strength | Baseline, 3 & 6 months
Serum phosphate | baselibe, 3 & 6 months
Feeling thermometer | Baseline, 3 & 6 months
Timed up and go | baseline, 3 & 6 months
Falls | continuous
Pulse wave velocity | baseline, 3 & 6 months
Bioimpedance | Baseline, 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ben Bull, Principal Investigator — Sir Charles Gairdner Hospital; Neil Boudville, Study Director — Sir Charles Gairdner Hospital
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia